CLINICAL TRIAL: NCT00463645
Title: An Open, Mono-Centre Trial to Investigate the Correlation Between the Interstitial and Arterial Blood Concentrations of Glucose During Subcutaneous Glucose Monitoring in Patients With Severe Sepsis at the Medical Intensive Care Unit
Brief Title: Investigation of Correlation Between Interstitial and Arterial Blood Glucose Concentrations in Septic Patients
Status: Completed | Type: Observational
Sponsor: Medical University of Graz (Other)
Other Study IDs: CM3_adipose
Record Dates: First submitted 2007-04-19; First posted 2007-04-20 (Estimated); Last update posted 2007-06-06 (Estimated); Status verified 2007-04

CONDITIONS: Severe Sepsis
MeSH Terms: conditions — Sepsis | interventions — Microdialysis

STUDY DESIGN:
Observational Model: Defined Population | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Procedure: microdialysis
Procedure: microperfusion

SUMMARY:
This is a mono-centre trial performed at the medical ICU at the Medical University Graz. There will be a study visit (V1) and a follow-up assessment (V2). In the study visit (V1) arterial blood glucose values will be monitored and subcutaneous sampling of interstitial fluid (ISF) with microdialysis for glucose determination and with microperfusion for cytokine-measurement will be performed. The study visit will last for 26 hours starting with the insertion of two catheters in the abdominal subcutaneous tissue (one microdialysis- and one microperfusion catheter). The primary hypothesis of the study is: Interstitial fluid glucose concentration profiles correlates to the arterial blood glucose concentration profile in patients with severe sepsis in the medical ICU.

ELIGIBILITY:
Inclusion Criteria:

* Patients in the medical ICU fulfilling criteria for severe sepsis
* Mechanical ventilation
* Increased blood glucose levels ( > 120 mg/dL; > 6.7 mM), or requiring insulin treatment.
* Age of patients in the range from 18 to 90 years.

Exclusion Criteria:

* Any disease or condition which the Investigator or the treating physician feels would interfere with the trial or the safety of the patient

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10
Dates: Start 2005-09; Study Completion 2006-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Thomas R. Pieber, MD., Principal Investigator — Medical University of Graz
Locations (1):
- Medical University Graz, Graz, Styria, Austria